CLINICAL TRIAL: NCT01820949
Title: Safety and Effectiveness of a Patient Blood Management (PBM) Program in Surgical Patients
Acronym: PBM
Status: Completed | Type: Observational
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Collaborators: University Hospital Schleswig-Holstein (Other); University Hospital, Bonn (Other); University Hospital Muenster (Other); Vifor Pharma (Industry); B. Braun Melsungen AG (Industry); CSL Behring (Industry); Fresenius Kabi (Industry)
Responsible Party: Principal Investigator, Professor Kai Zacharowski, M.D., Ph.D., FRCA, Prof. Dr. Dr. Kai Zacharowski, Johann Wolfgang Goethe University Hospital
Other Study IDs: 380/12
Record Dates: First submitted 2013-03-19; First posted 2013-03-29 (Estimated); Last update posted 2015-09-07 (Estimated); Status verified 2015-09

CONDITIONS: Surgery
Keywords: patient blood management; patients safety

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Control cohort: Standard care before implementation (pre-implementation)
- PBM cohort: After implementation of PBM program (post-implementation)

SUMMARY:
This study will evaluate clinical outcome after the step-wise implementation of a Patient Blood Management (PBM) Program in surgical patients at 4 hospitals.

DETAILED DESCRIPTION:
A PBM program will be implemented stepwise in four University Hospitals, with the intention to optimize preoperative hemoglobin concentration of patients and to standardize transfusion practice within hemotherapy. The PBM program includes 1) an algorithm with the aim to correct preoperative anemia in elective surgery, 2) a strict indication for the transfusion of red blood cells defined by the "Cross-sectional Guidelines for Therapy with Blood Components and Plasma Derivatives" for all surgical patients, and 3) a perioperative checklist for different blood-sparing techniques (e.g. cell-saver, normothermia, reduced blood samples, point-of-care diagnostics for bedside coagulation management).

Primary endpoint: Safety of the use of PBM program will be determined by comparability of the composite outcome (in-hospital myocardial infarction, stroke, acute renal failure, death of any cause, pneumonia and sepsis until discharge from hospital) between patients treated after implementation and patients treated before implementation (control cohort) of the PBM program.

The primary composite endpoint defined as described above will be registered electronically by analysis of Diagnosis Related Groups (DRG) codes. The frequency of these events will be compared between PBM and control cohort stratified by center with a one-sided Mantel-Haenszel test in a non-inferiority setting with significance level of α=2.5% and a non-inferiority margin of 1% for the incidence of the composite endpoint.

ELIGIBILITY:
Inclusion Criteria:

* All non- ambulant, surgical, anesthetized patients (≥18 years)
* General Surgery, Cardiac Surgery, Thoracic Surgery, Trauma Surgery, Vascular Surgery, Urology, Gynecology, Otolaryngology, Neurosurgery, Crania-Maxillofacial Surgery

Exclusion Criteria:

* ambulant and all non-surgical anesthetic procedures
* Surgery in the field of Dermatology or Ophthalmology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all surgical patients over a period of 24 months at 4 hospitals
Sampling Method: Non-Probability Sample
Enrollment: 110000 (Actual)
Dates: Start 2013-01; Primary Completion 2015-07 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Myocardial infarction, stroke, acute renal failure, death of any cause, pneumonia and sepsisComposite outcome | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks
  Composite endpoint defined as in-hospital myocardial infarction, stroke, acute renal failure, death of any cause, pneumonia and sepsis until discharge from hospital

SECONDARY OUTCOMES:
Length of stay on the intensive care unit | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks
Total hospital stay | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks
Total number of red blood cell transfusions during hospital stay | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks
Consumption of coagulation factors | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kai Zacharowski, MD, PhD, FRCA, Study Chair — Goethe University; Patrick Meybohm, MD, Principal Investigator — Goethe University; Erhard Seifried, MD, Principal Investigator — German Red Cross Blood Service Baden-Württemberg-Hessen, Institute for Transfusion Medicine and Immunohematology of the Goethe University Hospital, Frankfurt; Eva Herrmann, Principal Investigator — Institute of Biostatistics and Mathematical Modeling, Goethe University Frankfurt
Locations (4):
- Germany (4):
  - University Hospital Bonn, Bonn
  - University Hospital Frankfurt, Frankfurt
  - University Hospital Schleswig-Holstein, Kiel
  - University Hospital Muenster, Münster

REFERENCES:
- [Derived] Ellermann I, Bueckmann A, Eveslage M, Buddendick H, Latal T, Niehoff D, Geissler RG, Hempel G, Kerkhoff A, Berdel WE, Roeder N, Van Aken HK, Zarbock A, Steinbicker AU. Treating Anemia in the Preanesthesia Assessment Clinic: Results of a Retrospective Evaluation. Anesth Analg. 2018 Nov;127(5):1202-1210. doi: 10.1213/ANE.0000000000003583. PMID 29944518
- [Derived] Meybohm P, Herrmann E, Steinbicker AU, Wittmann M, Gruenewald M, Fischer D, Baumgarten G, Renner J, Van Aken HK, Weber CF, Mueller MM, Geisen C, Rey J, Bon D, Hintereder G, Choorapoikayil S, Oldenburg J, Brockmann C, Geissler RG, Seifried E, Zacharowski K; PBM-study Collaborators. Patient Blood Management is Associated With a Substantial Reduction of Red Blood Cell Utilization and Safe for Patient's Outcome: A Prospective, Multicenter Cohort Study With a Noninferiority Design. Ann Surg. 2016 Aug;264(2):203-11. doi: 10.1097/SLA.0000000000001747. PMID 27163948
- [Derived] Meybohm P, Fischer DP, Geisen C, Muller MM, Weber CF, Herrmann E, Steffen B, Seifried E, Zacharowski K; German PBM Study Core Group. Safety and effectiveness of a Patient Blood Management (PBM) program in surgical patients--the study design for a multi-centre prospective epidemiologic non-inferiority trial. BMC Health Serv Res. 2014 Nov 19;14:576. doi: 10.1186/s12913-014-0576-3. PMID 25927460
- See also: Safety and effectiveness of a Patient Blood Management (PBM) program in surgical patients - the study design for a multi-centre prospective epidemiologic non-inferiority trial — http://www.biomedcentral.com/content/pdf/s12913-014-0576-3.pdf